CLINICAL TRIAL: NCT00584675
Title: Nasopharyngeal 24 Hour pH Monitoring in Health Adult Volunteers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was never received so no patients were enrolled.
Sponsor: University of California, Davis (Other)
Responsible Party: Peter Belafsky, MD, Ph.D., University of California Davis
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 200714988-1
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; laryngopharyngeal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dx-pH Measurement Probe — Dx-pH Measurement Probe measures gaseous pH values in the nasopharynx and oropharynx over a period of 24 hours.

SUMMARY:
Involves a 24-hour pH probe study using the Dx-pH Measurement System on patients who do not have symptoms of laryngopharyngeal reflux or gastroesophageal reflux disease to establish normal values for the Dx-pH Measurement System.

DETAILED DESCRIPTION:
The specific aim of this study is to establish the normal range of values in an adult population with no symptoms of laryngopharyngeal reflux disease or gastroesophageal reflux disease using the Dx-pH Measurement System.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* no symptoms of laryngopharyngeal reflux or gastroesophageal reflux disease
* score less than 10 on Reflux Symptom Index

Exclusion Criteria:

* age less than 18
* known lidocaine allergy
* history of heartburn, regurgitation, chronic cough, voice changes, globus pharyngeus, excessive throat clearing, or swallowing problems
* score 10 or greater on Reflux Symptom Index
* current or past antacid use or other antireflux therapy
* history of antireflux surgery
* pregnancy
* current anticoagulation therapy (warfarin, heparin, aspirin, clopidogrel bisulfate)
* special/vulnerable populations (children, mentally handicapped, pregnant women, fetuses, prisoners, cognitive impairment, life-threatening disease, social or economic disadvantage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Estimated); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
To develop a range of normal values in adults without symptoms of laryngopharyngeal reflux. | At completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States